CLINICAL TRIAL: NCT01269580
Title: The Diabetic Foot: Relevance of Vascular Progenitor Cells as a Prognostic Marker of Cardiovascular Mortality, Restenosis, and Atherosclerotic Disease Progression in Treated Limb.
Brief Title: Diabetic Foot and Vascular Progenitor Cells
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Sponsor
Other Study IDs: 20/2008_Cardiovascolare
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes; Critical Limb Ischemia
MeSH Terms: conditions — Diabetes Mellitus; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic: Adult diabetic patients type 1 or 2, with chronic critical ischemia as defined by TASC 2007 criteria
- Not diabetic: Adult not diabetic with chronic critical ischemia

SUMMARY:
Type of Study: Pilot Study monocenter Study Duration: 18 months Subject Participation Duration: The patients are enrolled for the time of the blood withdrawl.

Follow up visit will be after 12 months from the enrollement.

Objectives:

The project will have two major objectives:

A)To validate the prognostic value of vascular progenitor cells, identified by flow cytometric analysis of antigenic phenotype, in a cohort of 109 patients with type-2 diabetes complicated by ischemic foot ulcers. Events are: cardiovascular mortality, major amputation, post-angioplasty restenosis , and development of new atherosclerotic plaques in treated limb B)To determine the mechanisms responsible for vascular progenitor cell dysfunction in the perspective of new therapies for the cure of the diabetic foot.

DETAILED DESCRIPTION:
This collaborative project aims to produce significant outputs for the identification of patients requiring intensification of therapy. Furthermore, the project will fill the gap in current knowledge on the post-genomic alterations that render diabetic vascular progenitor cells dysfunctional. In perspective, this might help us to design new therapies for the cure of the diabetic foot, including but not limited to stem cell therapy.

Primary Objectives:

To validate the prognostic value of vascular progenitor cells, identified by flow cytometric analysis of antigenic phenotype, in a cohort of 109 patients with type-2 diabetes complicated by ischemic foot ulcers.

Events are:

Cardiovascular mortality Major amputation Post-angioplasty restenosis Development of new atherosclerotic plaques in treated limb (follow up: 12 months).

Secondary Objectives:

To determine the mechanisms responsible for vascular progenitor cell dysfunction in the perspective of new therapies for the cure of the diabetic foot.

All the Units will contribute to the primary objective (to validate the prognostic value of vascular progenitor cells, identified by flow cytometric analysis of antigenic phenotype, in a cohort of 100 patients with type-2 diabetes complicated by ischemic foot ulcers). Furthermore, each Unit will focus on specific mechanistic targets, according to pilot data collected in previous and ongoing projects.

Dr Faglia, Head of the Diabetology Unit, Diabetic Foot Centre (IRCCS Multimedica-MM), will conduct the selection and enrollement of the patients, and collect all the clinical data for the study at the 12 month follow up visit.

The Unit leaded by Prof. Madeddu (IRCCS Multimedica), will perform the antigenic characterization of the vascular progenitor cells by flow cytometry, and conduct the migration assays.

The Unit leaded by Prof. Madeddu (IRCCS Multimedica)and the Unit leaded by Dr. Gaetano and Martelli (IDI, Rome) will be engaged with determining whether vascular progenitor cells dysfunction is mediated by specific epigenetic modifications. Epigenetics refers to the covalent modifications found in chromatin, on both the DNA and the accompanying histone proteins.

The Unit of Dr. Germani (IDI, Rome) will be focused on identification of growth factors, chemokines and cytokines in the serum of diabetic patients that could be involved in the deregulation of progenitor functions.

Since normal criteria are not already available, to conduct the analyses performed by the UO IDI, we need to enrol a group of 30 not-diabetic subjects age- and sex-matched to identify key changes to analyze in the entire group of patients.

Thirty patients coming to MM, UO Vascular Surgery, Dr Losa, for varicose vein treatment or carotid stenosis will be enrolled and subjected to blood withdrawal as described for the diabetic patients group.

Subject Inclusion Criteria:

Adult diabetic patients type 1 or 2, both men and women, with chronic critical ischemia as defined by TASC 2007 criteria (pain at rest, and/or ulcer or gangrene due to artheropaty: transcutaneous oximetry < 30 mmHg or pressure on the ankle < 70 mmHg).

Subject Exclusion Criteria:

* Cancer with adverse prognosis in months, or chemotherapic treatment
* Ongoing or planned pregnancy
* Lack of consent to participate to the study

Patients enrolment

At this time all patients will undergo all the following exams:

* General comprehensive visit (including: Chest RX, Rest ECG, and glycaemia plus glycosilated haemoglobin measurement)
* Ankle arterial pressure (Doppler cw measurement)
* Angiographyc study and angioplasty,if feasible, in the same time

IMPORTANT NOTE: At the enrolment visit and at follow up visit after 12 months will be performed:

* Ecodoppler
* Transcutaneous oximetry
* Completion of antigenic profiling
* Assessment of migratory capacity
* Characterization of major epigenetic signatures
* Paracrine profiling

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patients type 1 or 2
* Chronic critical ischemia as defined by TASC 2007 criteria (pain at rest, and/or ulcer or gangrene due to artheropaty: transcutaneous oximetry < 30 mmHg or pressure on the ankle < 70 mmHg)

Exclusion Criteria:

* Cancer with adverse prognosis in months, or chemotherapic treatment
* Ongoing or planned pregnancy
* Lack of consent to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with peripheral ischemia
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2009-02; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
post revascularization cardiovascualr mortality | 18 months

SECONDARY OUTCOMES:
post revascularization amputation | 18 months

OTHER OUTCOMES:
post revascularization restenosis | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Faglia, MD, Principal Investigator — IRCCS Multimedica
Locations (1):
- Diabetic Foot Center IRCCS MultiMedica, Sesto San Giovanni, Milan, Italy

REFERENCES:
- [Derived] Spinetti G, Specchia C, Fortunato O, Sangalli E, Clerici G, Caminiti M, Airoldi F, Losa S, Emanueli C, Faglia E, Madeddu P. Migratory activity of circulating mononuclear cells is associated with cardiovascular mortality in type 2 diabetic patients with critical limb ischemia. Diabetes Care. 2014 May;37(5):1410-7. doi: 10.2337/dc13-2084. Epub 2014 Feb 26. PMID 24574344